CLINICAL TRIAL: NCT02485665
Title: Efficacy of Personalized Extracorporeal Biofeedback Device for Pelvic Floor Muscle Training on Post-prostatectomy Incontinence
Brief Title: Efficacy of Extracorporeal Biofeedback Device for Post-prostatectomy Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Furun Medical (Industry)
Responsible Party: Principal Investigator, Seok-Soo Byun, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: L-2015-298
Record Dates: First submitted 2015-06-26; First posted 2015-06-30 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Prostate Neoplasm; Prostatectomy; Surgical Procedures, Robotic; Urinary Incontinence; Biofeedback; Pelvic Floor; Exercise
Keywords: Prostate cancer; Robot-assisted laparoscopic surgery; Radical prostatectomy; Post-prostatectomy incontinence; Pelvic floor muscle exercise; Extracorporeal biofeedback device
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Incontinence; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Kegel exercise education (No Intervention): Prostate cancer patients of control group will received Kegel exercise education for pelvic floor muscle exercise (PFME) to improve the post-prostatectomy incontinence after robot-assisted laparoscopic radical prostatectomy.
- Extracorporeal biofeedback device (Experimental): Prostate cancer patients of intervention group will received extracorporeal biofeedback device (Any Kegel) for pelvic floor muscle exercise (PFME) to improve the post-prostatectomy incontinence after robot-assisted laparoscopic radical prostatectomy.
  Interventions: Device: Extracorporeal biofeedback device (Any Kegel)

INTERVENTIONS:
Device: Extracorporeal biofeedback device (Any Kegel) — Prostate cancer patients of intervention group will received extracorporeal biofeedback device (Any Kegel) for pelvic floor muscle exercise (PFME) to improve the post-prostatectomy incontinence after robot-assisted laparoscopic radical prostatectomy. Enrolled patients in intervention group should be performed PFME regularly, based on following protocols: total exercise time (10 minutes/day), intensity (1.2 kgf), tension duration (10 sec/ 1 contraction), total exercise number (4 times/day)
  Arms: Extracorporeal biofeedback device

SUMMARY:
To evaluate the efficacy of postoperative pelvic floor muscle training using personalized extracorporeal biofeedback device among patients with post-prostatectomy incontinence

DETAILED DESCRIPTION:
* Post prostatectomy urinary incontinence (PPI) was common complication after radical prostatectomy among prostate cancer patients.
* The prevalence of post-prostatectomy urinary incontinence was reported at 87%.
* The pelvic floor muscle therapy (PFMT) using Kegel exercise was first methods to prevent PPI after prostatectomy.
* However, there was no standardized protocol of the PFMT and it was necessary of biofeedback to PFMT.
* Therefore, we hypothesis the efficacy of personalized device of PFMT with biofeedback among patients who underwent radical prostatectomy
* In this study, we evaluate the efficacy of postoperative pelvic floor muscle training using personalized extracorporeal biofeedback device among patients with post-prostatectomy incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer patients who underwent robotic radical prostatectomy
* Neurovascular saving at least one side
* Bladder neck reconstruction at prostatectomy
* Posterior reconstruction at prostatectomy
* Patients who have post-prostatectomy incontinence after Foley catheter removal

Exclusion Criteria:

* Patients who have not post-prostatectomy incontinence after Foley catheter removal
* Neurological deficits
* Anatomic deformities of pelvic bone
* Pelvic irradiation history
* History of other major urological procedures
* Complications influencing urinary incontinence

Ages: 20 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-03 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Recovery of urinary continence | postoperative 1 month
  weight of pad (g) by 24 hours pad test

SECONDARY OUTCOMES:
Recovery of urinary continence | postoperative 3 month
  weight of pad (g) by 24 hours pad test
Recovery of urinary continence | postoperative 1 and 3 months
  number of pads for 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Seok-Soo Byun, M.D.,Ph.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongam City, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Oh JJ, Kim JK, Lee H, Lee S, Jin Jeong S, Kyu Hong S, Eun Lee S, Byun SS. Effect of personalized extracorporeal biofeedback device for pelvic floor muscle training on urinary incontinence after robot-assisted radical prostatectomy: A randomized controlled trial. Neurourol Urodyn. 2020 Feb;39(2):674-681. doi: 10.1002/nau.24247. Epub 2019 Dec 2. PMID 31793032